CLINICAL TRIAL: NCT02750930
Title: An Open-label Extension to Study 200952 to Evaluate the Long-term Safety, Tolerability and Pharmacodynamics of Albiglutide Liquid Drug Product in Subjects With Type 2 Diabetes Mellitus
Brief Title: Extension to Study 200952 to Evaluate the Long-term Safety, Tolerability and Pharmacodynamics of Albiglutide Liquid Drug Product in Type 2 Diabetes Mellitus Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The termination was result of GSK business considerations and not due to quality, safety or efficacy concerns with any albiglutide formulations or study conduct
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204682
Record Dates: First submitted 2016-04-14; First posted 2016-04-26 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Extension; Long-term Safety; Pharmacodynamics; Albiglutide; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albiglutide arm (Experimental): Subjects will receive 50 milligrams (mg) albiglutide liquid drug product once weekly via auto-injector for 26 weeks.
  Interventions: Drug: Albiglutide; Device: Auto-injector

INTERVENTIONS:
Drug: Albiglutide — Albiglutide liquid drug product is provided as a fixed-dose, disposable auto-injector containing albiglutide liquid drug product (50 mg). Subjects will receive albiglutide 50 mg through subcutaneous injection in the abdomen, thigh or upper arm region via auto-injector. Albiglutide is a glucagon-like peptide-1 agonist (GLP-1 agonist).
Device: Auto-injector — The auto-injector delivers the albiglutide liquid drug product in an injection volume of 1.0 mL for the 50 mg dose.

SUMMARY:
Albiglutide has been developed for the treatment of type 2 diabetes mellitus (T2DM) as an adjunct to diet and exercise, as monotherapy, or in combination with existing therapies and has been approved by the United States (US) Food and Drug Administration (FDA), the European Medicines Agency (EMA) and other regulatory agencies. This is a 26 week, open-label, single group, multicenter, extension study to Study 200952. This extension study will provide extended safety, tolerability and immunogenicity data for the albiglutide liquid drug product. This extension study will comprise 2 study periods: treatment (26 weeks) and post-treatment follow-up (8 weeks). A maximum of 300 subjects will be eligible to take part in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the 26 week Treatment Phase of Study 200952
* Male or female
* Able and willing to provide informed consent.

Exclusion Criteria:

* Subject meets one or more of the withdrawal stopping criteria at Visit 1 (Week 26)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (25):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Lomita, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Columbia, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Shavano Prk, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 participants with Diabetes Mellitus type II, were enrolled in the study from 3 centres in United States of America. The study was conducted from 07 October 2016 to 21 March 2017. The study was terminated prematurely as a reflection of GlaxoSmithKline business considerations.
Pre-assignment Details: The participants who completed study 200952 and who were eligible, were included in this open-label extension study 204682. This was an extension study, hence visit 1 of this study was also a last treatment visit of study 200952 (NCT02683746).
Groups:
- Albiglutide Liquid: The participants in this arm, self-administered, albiglutide liquid drug product 50 milligram (mg) at a volume of 1 millilitre (mL) as a single dose subcutaneous injection in the abdomen, thigh or upper arm region, once weekly, for 26-weeks. It was administered on the same day each week, anytime during the day without regards to meals. The first dose was self-administered by the participant in the supervision from clinic staff. All further doses of study treatment were self-administered by the participant.
Period: Overall Study
Arm/Group | Albiglutide Liquid
Started | 8
Completed | 0
Not Completed | 8
Not completed — Study closed/terminated | 8

BASELINE CHARACTERISTICS:
Groups:
- Albiglutide Liquid: The participants in this arm, self-administered, albiglutide liquid drug product 50 mg at a volume of 1 mL as a single dose subcutaneous injection in the abdomen, thigh or upper arm region, once weekly, for 26-weeks. It was administered on the same day each week, anytime during the day without regards to meals. The first dose was self-administered by the participant in the supervision from clinic staff. All further doses of study treatment were self-administered by the participant.
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 7
  American Indian or Alaskan native | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product whether or not it is considered drug related. This would include any side effect, injury, toxicity, sensitivity reaction, abnormal or worsening of a laboratory value, concurrent illness or sudden death. Pre-existing conditions that worsen during a study will be reported as AEs. SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect, or is associated with liver injury or impaired liver function. Number of participants who reported any AE or SAE during this extension study or who had ongoing AE or SAE from study 200952 have been presented.
Time Frame: Up to Week 34
Population: Safety Population comprised of all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Groups:
- Albiglutide Liquid: The participants in this arm, self-administered, albiglutide liquid drug product 50 mg at a volume of 1 mL, as a single dose subcutaneous injection in the abdomen, thigh or upper arm region, once weekly, for 26-weeks. It was administered on the same day each week, anytime during the day without regards to meals. The first dose was self-administered by the participant in the supervision from clinic staff. All further doses of study treatment were self-administered by the participant.
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Participants
  Any SAE | 0
  Any AE | 2

2. Primary Outcome: Number of Participants With Physical Examination Abnormalities
Description: A full physical examination was planned to be done, at a minimum, assessment of the skin (including injection site), head, eyes, ears, nose, throat, thyroid, respiratory system cardiovascular system, abdomen (liver and spleen), lymph nodes, central nervous system and extremities was planned. The evaluation of skin (including injection site), respiratory system, cardiovascular system, abdomen (liver, spleen), and central nervous system was planned; however, it was not performed due to early termination of the study.
Time Frame: Up to Week 34
Population: Safety Population.
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Hematology Values of Potential Clinical Importance (PCI)
Description: Blood samples were collected from the participants to evaluate the hematology paramaters. The following hematology parameters were measured: platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), white blood cell (WBC) count, neutrophils, lymphocytes, monocytes, eosinophils, and basophils, at the specified timepoints (Week 0, 4, 10, 22, 26 and Week 34). Number of participants with hematology paramaters with PCI values has been reported.
Time Frame: Up to Week 34
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Participants | 1

4. Primary Outcome: Number of Participants With Clinical Chemistry Parameters of PCI
Description: The following clinical chemistry parameters were measured: blood urea nitrogen (BUN), creatinine, calcium, bicarbonate, potassium, sodium, chloride, uric acid, aspartate amino transferase (AST), alanine amino transferase (ALT), alkaline phosphatase, gamma glutamyl transferase (GGT), total and direct bilirubin, total protein, and albumin at the specified timepoints (Week 0, 4, 10, 22, 26 and Week 34). Number of participants with clinical chemistry paramaters with PCI values has been reported.
Time Frame: Up to Week 34
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Participants | 1

5. Primary Outcome: Number of Participants With Clinically Significant Urinalysis Abnormalities by Dipstick Method
Description: Urine samples were collected early morning from the participants at specified timepoints (Weeks 26 to 52). The following urinalysis parameters were measured: specific gravity, power of hydrogen (pH), glucose, protein, blood and ketones by dipstick; microscopic examination (if blood or protein was abnormal). Number of participants with no clinically significant abnormalities in urinalysis dipstick results were reported.
Time Frame: Up to 26 weeks
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Participants | 0

6. Primary Outcome: Number of Participants With Pulse Rate Values of PCI
Description: The pulse rate, was measured after completion of the electrocardiogram (ECG) sampling at specified timepoints (Week 0, 4, 10, 22, 26 and Week 34). The participants were asked to be either in semi-recumbent or sitting position. During blood withdraws the vitals were performed prior to blood collection. Number of participants with pulse rate values of PCI has been reported.
Time Frame: Up to Week 34
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Participants | 0

7. Primary Outcome: Number of Participants With Systolic and Diastolic Blood Pressure of PCI
Description: The systolic and diastolic blood pressure, were measured after completion of the ECG sampling at specified timepoints (Week 0, 4, 10, 22, 26 and Week 34). The participants were asked to be either in semi-recumbent or sitting position. During blood withdraws the vitals were performed prior to blood collection. Number of participants with systolic and diastolic blood pressure values of PCI has been reported.
Time Frame: Up to Week 34
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Participants | 0

8. Primary Outcome: Number of Participants With Clinically Significant Findings for 12-lead ECG
Description: A single 12-lead ECG was performed at the specified timepoints (Weeks 0, 26 and 34) during the study where the participant was instructed to be in semi-recumbent position for 10 to 15 minutes before obtaining the ECG. An ECG machine that automatically calculated the heart rate and measures like the PR, QRS, QT, and corrected QT intervals. Number of participants with clinically significant findings in ECG results has been reported.
Time Frame: Up to Week 34
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 8
Participants | 0

9. Primary Outcome: Number of Participant With Positive Results of Anti-albiglutide Antibody Production Over Time
Description: Anti-albiglutide antibodies were planned to be assessed using a validated enzyme-linked immunosorbent assay, which utilized a tiered testing approach. It was to be collected at specified timepoints at Week 0, Week 4, Week 10, Week 26 and Week 34 (follow-up). Confirmed positive samples were to be titrated to obtain the titer of anti-albiglutide antibodies. The number of participants with positive results of anti-albiglutide antibody production was to be reported. However, due to early termination only limited number of key safety data was analyzed. This study 204682 was planned as an extension of the main study, 200952 and was supposed to end well after the main study. However, the 204682 extension study was terminated prior to completion of the main study 200952, which is a double-blind study. To preserve the integrity of the main study 200952, results of anti-albiglutide antibody were not completed after the termination.
Time Frame: Up to Week 34
Population: Safety population.
Arm/Group | Albiglutide Liquid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment (Week 1 of this extension study) to upto follow-up (Up to Week 34)
Description: Safety population was used. On treatment AEs and SAEs were reported.
Arm/Group | Albiglutide Liquid
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide Liquid (N=8)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Tooth abscess (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT02750930/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT02750930/SAP_001.pdf